CLINICAL TRIAL: NCT06347224
Title: Navigating the Both Column Fixation Corridor: Anatomical Insights From a Virtual Pelvic Screw Placement Study
Brief Title: Both Column Fixation Corridor in Pelvic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Vedat Öztürk, Specialist Doctor in Orthopedics and Traumatology, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: BCFC-BCS-VIRTUAL2024
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Acetabular Fractures
Keywords: both column screw; percutaneous fixation; acetabulum

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- male group (Other): Male Group: In this study, the male group consists of 200 healthy adult men selected from hospital radiology archive records, who have undergone pelvic computed tomography (CT) scans for various reasons. These individuals were chosen excluding those with pelvic fractures, anatomical abnormalities, or severe osteoporosis. The age range of the male group is between 18 and 65 years, with a median age of approximately 39.4 years. Analyses conducted on the male group focus on concepts such as the Both Column Fixation Corridor (BCFC) and Both Column Screws (BCS), evaluating the feasibility, gender-specific anatomical differences, and potential advantages of this new fixation technique.
  Interventions: Procedure: Virtual placement of lag screws in both columns of the acetabulum on 3D pelvic CT models.
- female group (Other): Female Group: Similarly, the female group comprises 200 healthy adult women who have had pelvic CT scans for any reason, selected from hospital radiology archives. Like the male group, these individuals meet the specific criteria set for the study. The age range for the female group is also between 18 and 65 years, with a median age comparable to that of the male group. The analysis of the female group centers on the feasibility of applying BCFC and BCS, taking into account the unique anatomical structures of the female pelvis and their implications for surgical planning. The work on this group aims to enhance the understanding of gender-specific anatomical variations and integrate this knowledge into surgical practices.
  Interventions: Procedure: Virtual placement of lag screws in both columns of the acetabulum on 3D pelvic CT models.

INTERVENTIONS:
Procedure: Virtual placement of lag screws in both columns of the acetabulum on 3D pelvic CT models. — The intervention aims to simulate a percutaneous fixation technique that could be applied in a real surgical environment, offering insights into the potential for personalized surgical planning and optimization of outcomes for patients with acetabular fractures. This virtual approach allows for the exploration of various screw placement strategies without the ethical and practical constraints of direct clinical experimentation.

SUMMARY:
The concepts of the Both Column Fixation Corridor (BCFC) and Both Column Screws (BCS) have emerged as innovative approaches in orthopedic surgery yet have not been extensively explored in the literature. This study aims to evaluate the feasibility and potential advantages of this novel screw fixation technique, thereby filling the existing gap in knowledge and establishing standards for its application.

DETAILED DESCRIPTION:
Pelvic CT data will be collected from 400 healthy adults, including 200 males and 200 females. The Synapse software will be utilized to simulate the placement of both anterior and posterior Both Column Screws (BCS) in the Both Column Fixation Corridor (BCFC). Screws will be virtually implanted into the BCFC using the "Ozturk Procedure," a technique developed based on clinical practice. Measurements will include the thickness and length of each BCS for both anterior (aBCS) and posterior (pBCS) placements, as well as the distances from the screw centers to the spina iliaca anterior superior (SIAS). Additionally, the necessary caudo-cranial (CCT) and centro-lateral tilts (CLT) for achieving axial fluoroscopic visualization of the BCFC will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Both male and female participants.
* Participants with healthy pelvic anatomy as determined by CT imaging, without any previous fractures, deformities, or surgical interventions that could alter the pelvic structure.

Exclusion Criteria:

* History of pelvic or acetabular fractures.
* Previous pelvic surgeries that could alter the anatomical structure.
* Conditions significantly affecting bone quality, such as osteoporosis or metabolic bone diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Successful Visualization of Both Column Fixation Corridor (BCFC) and Placement of Both Column Screws (BCS) | up to 3 months
  This measure evaluates whether the axial fluoroscopic image of the BCFC can be successfully demonstrated across all participant populations, regardless of gender, and whether it's feasible to place two BCS within the BCFC, one anterior and one posterior, in the surgical treatment of pelvic and acetabular fractures. It also examines gender-specific anatomical variations associated with the BCFC and BCS and their implications for surgical planning.

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Öztürk, Dr., Principal Investigator — Bakırköy Dr. Sadi Konuk Education and Research Hospital, Department of Orthopedics and Traumatology
Locations (1):
- Bakırköy Dr. Sadi Konuk Education and Research Hospital, Department of Orthopedics and Traumatology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) from this study is in place. Due to the sensitivity of the data and the need to protect participant confidentiality, these data will be accessible only to the research team and will not be shared with any third parties.

REFERENCES:
- [Background] Ozturk V, Celik M, Koluman AC, Duramaz A, Kural C, Bilgili MG. Fluroscopy-assisted transiliac antegrade lag screw placement technique in both columns of acetabulum: A novel procedure. Orthop Traumatol Surg Res. 2024 Sep;110(5):103872. doi: 10.1016/j.otsr.2024.103872. Epub 2024 Mar 26. PMID 38548224